CLINICAL TRIAL: NCT02014337
Title: Phase 1 Study of Mifepristone in Combination With Eribulin in Patients With Locally Advanced/Metastatic Breast or Other Specified Solid Tumors, With a Dose Expansion Cohort in Patients With Triple Negative Breast Cancer.
Brief Title: Mifepristone and Eribulin in Patients With Metastatic Triple Negative Breast Cancer or Other Specified Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1073-500
Record Dates: First submitted 2013-12-04; First posted 2013-12-18 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer; Ovarian Epithelial Cancer Recurrent; Sarcoma; Non-small Cell Lung Cancer; Carcinoma, Transitional Cell; Prostate Cancer; Prostatic Neoplasms
Keywords: Mifepristone; Eribulin Mesylate; Breast Cancer; Ovarian Cancer; Sarcoma; Non-small cell lung cancer; Carcinoma, transitional cell; Prostate cancer; Prostatic neoplasms
MeSH Terms: conditions — Breast Neoplasms; Sarcoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell; Prostatic Neoplasms; Ovarian Neoplasms | interventions — Mifepristone; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mifepristone and Eribulin in combination (Experimental): Single Arm
  Interventions: Drug: Mifepristone and Eribulin in combination

INTERVENTIONS:
Drug: Mifepristone and Eribulin in combination — Single Arm, Two Parts Part 1: Dose Escalation Phase to determine MTD and RP2D in up to 20 patients Part 2: Dose Expansion Phase at RP2D in 20 patients
  Other Names: Korlym®; Halaven

SUMMARY:
This is a study to assess the safety of the combination of mifepristone and eribulin in patients with metastatic or locally advanced unresectable breast or other specified solid tumors, and determine preliminary efficacy of the combination of mifepristone and eribulin in patients with metastatic or locally advanced unresectable Triple Negative Breast Cancer (TNBC). The structure for the study is a single arm, non-randomized, open-label, multicenter trial with no control group. The study will be conducted at up to 11 sites, with up to 40 evaluable patients

DETAILED DESCRIPTION:
There will be two parts to the study: Part 1, a dose escalation phase, in which the MTD and RP2D will be determined in up to 20 patients with metastatic breast or other specified solid tumors, regardless of receptor status; and Part 2, a dose expansion phase in which a preliminary estimate of efficacy will be made in an expansion group of up to 20 patients with glucocorticoid receptor-positive metastatic TNBC at the RP2D.

Treatment will be administered in 21-day cycles, with the exception of the first cycle, which will be of 28 days duration with a lead-in of 7 days dosing of mifepristone.

Cycle 1 (28-day cycle): Mifepristone administered orally (PO) with food once daily for 28 days. Eribulin will be administered intravenously (IV) over 2 to 5 minutes on days 8 and 15.

Cycle 2 and beyond (21-day cycle): Mifepristone administered orally (PO) with food once daily for 21 days. Eribulin will be administered intravenously (IV) over 2 to 5 minutes on days 1 and 8.

Enrollment in Part 2 of the study (dose expansion) will occur once the RP2D has been determined. Patients in the dose expansion study must have TNBC disease that is glucocorticoid receptor-positive (by immunohistochemistry [IHC]). Patients will be treated in repeated 21-day cycles until progression or another withdrawal criterion is met.

Part 1 of the study is complete. Part 2 of the study is ongoing.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent given prior to study-specific screening procedures
2. ≥ 18 years old

Part 2, dose expansion:

1. Diagnosis of TNBC: < 1% cells positive for ER/progesterone receptor, and HER2 IHC score of 0 or 1, or FISH HER2+ ratio of less than 1.8; patients with low ER IHC (> 1% but < 10% cells positive), but negative by genomic assay are eligible
2. Inoperable metastatic or locally advanced unresectable disease
3. Patients should have received a minimum of one, and up to five prior chemotherapy regimens
4. Must have submitted a diagnostic FFPE tumor tissue sample to confirm tumor GR positivity. Tumor tissue may be from primary or metastatic lesion. In the absence of sufficient tissue to complete IHC, a tumor biopsy will be required.
5. Tumor must be glucocorticoid receptor positive TNBC (≥10% positive cells by IHC of tumor biopsy)
6. Must have measurable disease (RECIST v1.1) in at least one lesion not previously irradiated unless documented evidence of progression
7. Patients with treated, stable brain metastases eligible providing treatment was ≥4 weeks prior to initiation of study drug, and baseline CT or MRI negative for new brain metastases. Must not require therapy with corticosteroids.
8. ECOG performance status 0 or 1
9. Must have adequate bone marrow and renal/hepatic function at the screening visit (≤7 days preceding the lab assessment):

   i. ANC ≥ 1,500/mm3, without G-CSF

   ii. Platelets ≥ 100,000/mm3, without transfusion

   iii. Hemoglobin ≥ 9 g/dL, without transfusion support

   iv. AST or ALT ≤ 3 × ULN

   v. Total serum bilirubin ≤ 1.5 times ULN

   vi. Serum creatinine ≤ ULN

   vii. Potassium and magnesium levels within normal limits. If below the lower limit of normal, must have levels corrected by supplementation prior to starting study drug.

   viii. albumin > 3.0 g/dL
10. PT/aPIT ≤ 1.5 x ULN
11. Disease-free period of > 3 years from any other previous malignancies, excluding curatively treated basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix.
12. Female patients of childbearing potential must have a negative serum pregnancy test. Sexually active patients must be willing to use non-hormonal contraception, including condom use by male partner, and barrier method by the female partner during the treatment period and for at least 3 months after the last dose of the study drug. Females considered not of childbearing potential include those who have been in menopause > 2 years, or are surgically sterile (status post tubal ligation or hysterectomy).
13. Must be able and willing to comply with the study visit schedule and study procedures.
14. Able to take oral medications

Exclusion Criteria:

1. Systemic cytotoxic therapies or radiotherapy ≤14 days prior to day 1 cycle 1
2. Major surgery within 4 weeks, or minor surgery within 2 weeks prior to day 1 of cycle 1
3. Endometrial bleeding
4. For two weeks prior to day 1 cycle 1, administration of specified cytochrome P450 3A (CYP3A) inducers
5. Patients who are taking simvastatin or lovastatin. Patients should be switched to alternative therapies a minimum of 2 weeks before starting study drug
6. Patients who have been treated with an investigational agent <21 days prior to day 1 of cycle 1
7. Concomitant use of biological agents including growth factors. Exception: 3- to 6-patient breast cancer cohort enrolled to explore the use of prophylactic growth-factor support of a 1.4 mg/m2 dose of eribulin.
8. Patients who require treatment with systemic corticosteroids for serious medical conditions or illnesses (e.g. immunosuppression after organ transplantation)
9. History of significant cardiac disease. Includes second/third degree heart block; significant ischemic heart disease; mean QTc interval > 480 msec prior to study start; poorly controlled hypertension; congestive heart failure of NYHA Class II or worse
10. Pregnant or breast-feeding
11. Any other significant co-morbid conditions that would impair study participation or cooperation
12. In Part 2, unable or unwilling to consent to provision of tumor tissue for GR assay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Determine the MTD and recommended Phase 2 dose (RP2D) of the combination of mifepristone and eribulin in patients with metastatic or locally advanced unresectable breast or other specified solid tumors. | 28 days
  In the dose escalation phase: MTD time frame is within 28 days of first dose (Cycle 1)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Nanda, MD, Principal Investigator — University of Chicago
Locations (11):
- United States (11):
  - ACRC/Arizona Clinical Research Center Inc., Tucson, Arizona
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Rita Nanda, MD, Chicago, Illinois
  - Quest Research, Royal Oaks, Michigan
  - St. Luke's Cancer Institute, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No